CLINICAL TRIAL: NCT00001301
Title: Chronic and Late Effects of Non-Hodgkin's Lymphoma and Its Treatment in Long Term Survivors
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920242; 92-C-0242
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Adverse Effects; Burkitt's Lymphoma; Diffuse Large Cell Lymphoma; Extended Remission; Health Status; Lymphoblastic Lymphoma; Molecular Studies
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Precursor Cell Lymphoblastic Leukemia-Lymphoma

SUMMARY:
Non-Hodgkin's lymphoma has been studied in the Pediatric Branch for at least 20 years, during which time a number of different treatment protocols have been used. Approximately 110 patients have apparently been cured of their lymphoma. The present protocol has no therapeutic component, but is designed to document the late effects that may have been encountered by our patients, either as a consequence of the disease or its treatment. In essence, patients who consent to participate will be asked a series of questions pertaining to the quality of their life and possible medical problems that they may be encountering. In addition, they will receive a complete physical examination and undergo non-invasive investigations designed to identify the presence of unsuspected late effects. Investigators in the Eye Clinic, Dental Clinic, Audiology, Cardiology and Endocrinology departments will participate in the protocol. As a part of the study, blood samples will be obtained to investigate the possibility that predisposing genetic factors may be identifiable in the patients normal cells (e.g., p53 mutations, evidence of DNA instability). If such abnormalities are detected, blood samples from family members will also be examined to determine whether the defect was inherited.

DETAILED DESCRIPTION:
Non-Hodgkin's lymphoma has been studied in the Pediatric Branch for at least 20 years, during which time a number of different treatment protocols have been used. Approximately 110 patients have apparently been cured of their lymphoma. The present protocol has no therapeutic component, but is designed to document the late effects that may have been encountered by our patients, either as a consequence of the disease or its treatment. In essence, patients who consent to participate will be asked a series of questions pertaining to the quality of their life and possible medical problems that they may be encountering. In addition, they will receive a complete physical examination and undergo non-invasive investigations designed to identify the presence of unsuspected late effects. Investigators in the Eye Clinic, Dental Clinic, Audiology, Cardiology and Endocrinology departments will participate in the protocol. As a part of the study, blood samples will be obtained to investigate the possibility that predisposing genetic factors may be identifiable in the patients normal cells (e.g., p53 mutations, evidence of DNA instability). If such abnormalities are detected, blood samples from family members will also be examined to determine whether the defect was inherited.

ELIGIBILITY:
Patients with a histologic diagnosis of small noncleaved cell (undifferentiated) (SNCL), lymphoblastic (LL), and large cell lymphoma (LCL) who were treated according to National Cancer Institute Pediatric Branch non-Hodgkin's lymphoma protocols 74-0, 75-6, 76-5, 77-04, 85-C-67, and 89-C-41A, and who have been in continuous remission for one year or longer following completion of treatment.

Patients who have relapsed and been successfully re-treated are not excluded, except for patients with lymphoblastic lymphoma who have been re-treated according to acute lymphoblastic leukemia protocols.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107
Dates: Start 1992-08; Study Completion 2000-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ziegler JL, DeVita VT, Graw RG Jr, Herzig G, Leventhal BG, Levine AS, Pomeroy TC. Combined modality treatment of American Burkitt's lymphoma. Cancer. 1976 Dec;38(6):2225-31. doi: 10.1002/1097-0142(197612)38:63.0.co;2-f. PMID 1036716
- [Background] Appelbaum FR, Deisseroth AB, Graw RG Jr, Herzig GP, Levine AS, Magrath IT, Pizzo PA, Poplack DG, Ziegler JL. Prolonged complete remission following high dose chemotherapy of Burkitt's lymphoma in relapse. Cancer. 1978 Mar;41(3):1059-63. doi: 10.1002/1097-0142(197803)41:33.0.co;2-n. PMID 638947
- [Background] Magrath IT, Janus C, Edwards BK, Spiegel R, Jaffe ES, Berard CW, Miliauskas J, Morris K, Barnwell R. An effective therapy for both undifferentiated (including Burkitt's) lymphomas and lymphoblastic lymphomas in children and young adults. Blood. 1984 May;63(5):1102-11. PMID 6546890